CLINICAL TRIAL: NCT03391973
Title: A Multi-Centre, Single Arm, Phase 2 Trial of Pembrolizumab in Treatment Naïve Patients With Poor-Prognosis Carcinoma of Unknown Primary Site
Brief Title: Pembrolizumab in Patients With Poor-Prognosis Carcinoma of Unknown Primary Site (CUP)
Acronym: CUP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Tom Baker Cancer Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK-3475-418
Record Dates: First submitted 2017-11-06; First posted 2018-01-05 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Carcinoma of Unknown Primary
Keywords: CUP; Pembrolizumab; KEYTRUDA
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is a multi-centre, single arm phase 2 study of Pembrolizumab (Keytruda™ or MK-3475) in treatment naïve patients with poor prognosis carcinoma of unknown primary site (CUP).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Arm 1 - Pembrolizumab (Experimental): Arm 1 - Pembrolizumab injection dosed at 200 mg given Q3 weeks by IV infusion on Day 1 of each 3 week cycle.
  Interventions: Drug: Pembrolizumab Injection

INTERVENTIONS:
Drug: Pembrolizumab Injection — Pembrolizumab 200 mg will be administered as a 30 minute IV infusion Q3W.
  Other Names: Keytruda

SUMMARY:
Abbreviated Title: Pembrolizumab in Patients with Poor-Prognosis Carcinoma of Unknown Primary Site (CUP) Trial Phase: 2 Clinical Indication: Treatment naïve patients with poor prognosis carcinoma of unknown primary site Trial Type: Single arm phase 2 Type of control: Not applicable Route of administration: Intravenous Trial Blinding: Not applicable Treatment Groups: 1) Pembrolizumab 200 mg IV every 3 weeks for up to 24 months. Total Number of trial subjects:25 Estimated enrollment period: 24 months Estimated duration of trial: 48 months Duration of Participation: 24 months

DETAILED DESCRIPTION:
This is a multi-centre, single arm phase 2 study of Pembrolizumab (Keytruda™ or MK-3475) in treatment naïve patients with poor prognosis carcinoma of unknown primary site (CUP). Participants will receive Pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle for up to 24 months. Patients will be evaluated for response every 9 weeks. Patients with objective response to treatment and those with stable disease will continue to receive Pembrolizumab. Patients with tumor progression will be discontinued from the study. Patients with progressive disease (PD), but showing a clinical benefit, may continue on Pembrolizumab, as per the discretion of the responsible Qualified Investigator. Response will be evaluated as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically (or cytologically) documented, metastatic carcinoma with no primary site identified. The following tests are required to exclude a primary site of disease: complete history and physical examination, blood chemistry (including serum tumor marker for prostate-specific antigen (PSA) in men, alpha-fetoprotein (AFP), β-human chorionic gonadotropin (β-hCG)) and mammography in women, urinalysis, thoracic and abdominopelvic computed tomography scans, bone scan, and symptom or sign-oriented imaging or endoscopic studies).
2. Have adenocarcinoma, a poorly differentiated carcinoma, or any squamous cell carcinomas.
3. Be willing and able to provide written informed consent for this trial.
4. Be ≥ 18 years of age on day of signing informed consent.
5. Have documented measurable disease based on RECIST 1.1. via Computerized Tomography (CT) or Magnetic Resonance Imaging (MRI).
6. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 calendar days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived Formalin-Fixed, Paraffin-Embedded (FFPE) Block(s).
7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Must have a documented negative urine or serum pregnancy test within 7 days prior to receiving the first dose of study medication if female and of childbearing potential. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test is required.
9. Female subjects of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity from the time they sign the informed consent form prior to start of therapy through 120 calendar days after the last dose of study medication. Subjects of childbearing potential are defined as those who have not been surgically sterilized or have not been free from menses for > 1 year.
10. Male subjects must agree to use 2 adequate methods of contraception from the time they sign the informed consent form prior to start of therapy through 120 calendar days after the last dose of study therapy. Examples include: condoms, spermicidal jelly, and abstinence.
11. Demonstrate adequate organ function as defined in Table 1 below. All screening labs must be performed within 7 calendar days of treatment initiation.

Exclusion Criteria:

1. CUP suspected to be lymphomas (e.g. staining for leukocyte common antigen), malignant melanoma (e.g. staining for both S100 and HMB45), extragonadal germ cell neoplasms (e.g. staining for both AFP and β-hCG), sarcomas (e.g. staining for cytokeratins and vimentin), neuroendocrine tumors (e.g. staining for chromogranin and synaptophysin), and prostatic adenocarcinomas in men (e.g. staining for PSA).
2. Patient subgroups that are suitable for well-defined treatments: (e.g. women with adenocarcinoma involving axillary lymph nodes as the only site of disease, women with papillary serous carcinoma of the peritoneum, patients with squamous cell carcinoma that involved either cervical or inguinal lymph nodes only, patients with poorly differentiated carcinomas that suggested germinal tumors and with elevated levels of β-hCG and/or AFP, and patients with carcinoma that involved a single, potentially resectable site) also are excluded from enrollment.
3. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
4. Has a confirmed diagnosis of immunodeficiency or is receiving documented systemic steroid therapy or any other form of immunosuppressive therapy within 7 calendar days prior to the first dose of Pembrolizumab.
5. Has a known history of active Tuberculosis Bacillus (TB).
6. Hypersensitivity to Pembrolizumab or any of its excipients (L-histidine, L-histidine hydrochloride monohydrate, Sucrose or Polysorbate 80).
7. Has had radiation therapy within 14 calendar days prior to the first dose of treatment. If subject undergone radiation, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy as per the discretion of the Qualified Investigator.
8. Has had prior chemotherapy, targeted small molecule therapy, or prior anti-cancer mAb.
9. If subject has undergone major surgery, they must have recovered adequately from the complications from the surgery prior to starting therapy as per the discretion of the Qualified Investigator.
10. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
11. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by CT brain or MRI brain for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 calendar days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
12. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
13. Has a history of (non-infectious) pneumonitis or current pneumonitis.
14. Has an active infection requiring systemic therapy.
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating Qualified Investigator.
16. Has known psychiatric or substance abuse disorders that would interfere with compliance with the requirements of the trial.
17. Is pregnant or breastfeeding, or planning to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 calendar days after the last dose of trial treatment.
18. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
19. Has a known history of Human Immunodeficiency Virus (HIV).
20. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA is detected).
21. Has received a live vaccine within 30 calendar days of planned start of study therapy.
22. Has previous organ and/or bone marrow transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants that develop an objective response to treatment. | Within 3 years
  The objective response rate will be assessed by RECIST 1.1
Number of participants that develop an adverse event to treatment. | Within 3 years
  Treatment related adverse events will be assessed using CTCAE v4.0.

SECONDARY OUTCOMES:
The overall survival (OS) of participants. | Within 4 years
  OS is the time from treatment initiation to death due to any cause
The progression free survival (PFS) of participants. | Within 4 years
  Progression will be assessed by RECIST 1.1
The duration of response (DOR) of participants. | Within 4 years
  Response will be assessed by RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Jose Monzon, MD, Principal Investigator — Arthur J.E. Child Comprehensive Cancer Centre
Locations (3):
- Canada (3):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario